CLINICAL TRIAL: NCT02701439
Title: Small Membrane Filtration (SMF) Method to Improve the Performance of Smear Microscopy for the Diagnosis of Pulmonary Tuberculosis in a High HIV Prevalence Setting
Brief Title: SMF to Improve Performance of Microscopy for the Diagnosis of PTB in a High HIV Prevalence Setting
Acronym: PTB
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Boston University (Other); University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: SMF-01
Record Dates: First submitted 2013-02-16; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — TB isolates from sputum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV-infected: Enrollment of 740 HIV-infected adults with suspicion of pulmonary TB.
  Following the Ugandan National Tuberculosis and Leprosy Programme (NTLP) guidelines, all enrolled TB suspects will undergo the following standardized evaluation:
  * Abbreviated demographic and clinical evaluation
  * TB history and evaluation
  * Obtain three sputum samples - one early morning sample and two spot samples
  * HIV testing (and CD4 if positive)
  * Chest radiograph
  * Small membrane filtration intervention
  Interventions: Device: Small membrane filtration
- HIV negative: Enrollment of 350 HIV negative adults with suspicion of pulmonary TB.
  Following the Ugandan National Tuberculosis and Leprosy Programme (NTLP) guidelines, all enrolled TB suspects will undergo the following standardized evaluation:
  * Abbreviated demographic and clinical evaluation
  * TB history and evaluation
  * Obtain three sputum samples - one early morning sample and two spot samples
  * HIV testing (and CD4 if positive)
  * Chest radiograph
  * Small membrane filtration intervention
  Interventions: Device: Small membrane filtration

INTERVENTIONS:
Device: Small membrane filtration — Following the Ugandan National Tuberculosis and Leprosy Programme (NTLP) guidelines, all enrolled TB suspects will undergo the following standardized evaluation:
  * Abbreviated demographic and clinical evaluation
  * TB history and evaluation
  * Obtain three sputum samples - one early morning sample and two spot samples
  * HIV testing (and CD4 if positive)
  * Chest radiograph
  * Small membrane filtration intervention will be administered to both arms

SUMMARY:
This study is investigating a better method to see if someone has tuberculosis (TB) as compared to the method that is being used now.

DETAILED DESCRIPTION:
TB is a disease caused by a bacterium called Mycobacterium tuberculosis that can affect the lungs or other parts of the body. In most of the world and in Mbarara, Uganda, the method of diagnosis that is used is AFB smear microscopy. This method is widely available, inexpensive and rapid. However, this method's ability to truly detect people having TB is poor. That is, if someone has TB, the test results may say that they are negative, leading to delays in diagnosis, disease progression, and an ongoing transmission of the bacteria.

The new test for TB diagnosis we are studying is called the Small Membrane Filtration (SMF) method. This test that is being compared to the method currently being used and is very similar to the one that is currently used (standard smear microscopy) but has the advantage of concentrating the sputum (mucus) so that we can more easily see if bacteria are present in the sputum. It is hoped that a better way of knowing if someone has TB will help doctors decide when people need to be treated for TB and when not, which will improve the health of patients and help avoid passing the infection to others.

This study will enroll 740 HIV-infected and 310 HIV-uninfected adults with culture confirmed pulmonary TB. These individuals will be identified prospectively at two TB clinics in Mbarara, Uganda.

Study hypothesis: The investigators will assume that one sputum sample will be equivalent to two (null hypothesis) with respect to sensitivity unless we have evidence that the use of two has higher sensitivity (alternative hypothesis). The investigators will assume that SMF is equivalent to AFB smear with respect to sensitivity and specificity unless the investigators find evidence it is superior. The investigators will assume that SMF is equivalent to Xpert unless the investigators find evidence that Xpert is superior.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Pulmonary TB suspect defined as any person who presents with a productive cough for more than 2 weeks AND accompanied by at least one other respiratory symptom (shortness of breath, chest pains, hemoptysis) and/or constitutional symptom (loss of appetite, weight loss, fever, night sweats, and fatigue) (6).
* Willing to undergo TB evaluation and spontaneously expectorate ≥2 mL of sputum
* Willing to be tested for HIV, if no results available within past 6 months

Exclusion Criteria:

* Too ill or unable to provide written consent
* Treated with TB drugs for more than 3 days
* Extra-pulmonary or disseminated TB without pulmonary involvement (i.e. no cough)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a suspected diagnosis of pulmonary TB attending two TB clinics in Mbarara, Uganda
Sampling Method: Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of SMF method and Xpert MTB/RIF assay | 24 months
  The primary endpoints of this laboratory-based study will be to determine the sensitivity and specificity of the SMF method and Xpert MTB/RIF assay, using manual MGIT liquid culture as the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Yap Boum II, PhD, Principal Investigator — Epicentre
Locations (1):
- Epicentre Mbarara Research Base, Mbarara, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No